CLINICAL TRIAL: NCT03746808
Title: Development and Testing of a Just-in-Time Adaptive Smart Phone Intervention
Brief Title: Development and Testing of a Just-in-Time Adaptive Smart Phone Intervention to Reduce Drinking Among Homeless Adults
Acronym: Smart-T
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Texas Health Science Center (Other)
Collaborators: University of Oklahoma (Other)
Responsible Party: Principal Investigator, Scott Walters, PhD, Regents Professor, University of North Texas Health Science Center
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 1R34AA024584-01A1 (NIH)
Record Dates: First submitted 2018-11-13; First posted 2018-11-20 (Actual); Results first posted 2022-11-18 (Actual); Last update posted 2022-11-18 (Actual); Status verified 2022-11

CONDITIONS: Alcohol Use Disorder; Treatment; Homelessness
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EMA only (Placebo Comparator): Phase I will use smartphones and passive sensing to monitor geolocation, psychosocial variables (e.g., stress, urge to drink), and alcohol use in a group of 80 homeless adults with an AUD who are receiving shelter-based treatment.
  Interventions: Behavioral: EMA + App/Treatment Messages
- EMA + App/Treatment Messages (Active Comparator): Phase III will pilot test the newly developed app for utility, satisfaction, and preliminary effectiveness in a group of 40 homeless adults with an AUD who are receiving shelter-based treatment. The investigators will compare Phase III participants (i.e., received Metrocare, EMAs, and tailored treatment messages) to Phase I participants (i.e., received Metrocare and EMAs only) to examine the preliminary effectiveness of the app.
  Interventions: Behavioral: EMA + App/Treatment Messages

INTERVENTIONS:
Behavioral: EMA + App/Treatment Messages — This study will develop and test a "just-in-time" adaptive intervention to reduce alcohol use among homeless adults. Phase I will use smartphones and passive sensing to monitor geolocation, psychosocial variables (e.g., stress, urge to drink), and alcohol use in a group of 80 homeless adults with an AUD who are enrolled in shelter-based treatment. Phase II will use this information to create a risk algorithm and tailored treatment messages that anticipate and intervene to prevent alcohol use.

SUMMARY:
Homeless adults are 8 times as likely to be alcohol dependent compared with adults in the general population, yet few studies have examined the precipitants of alcohol use in this vulnerable population. Ecological momentary assessments (EMAs) that involve repeated assessment of thoughts/mood/behaviors (e.g., via smart phone) is currently the most accurate way to assess individuals in real-time in their natural environments. Advances in smartphone technology also allow for the collection of continuous geolocation and other passive sensing data. Thus, researchers can now link environmental risks and protective factors to outcomes, without reliance on subjective reporting alone. Building on prior work, this study will use a three-phase study to develop and test a "just in time" adaptive intervention to reduce alcohol use in homeless men and women. Phase I will use smartphones and passive sensing technologies to monitor geolocation, psychosocial variables (e.g., stress, affect, urge to drink), and alcohol use in a group of 80 homeless adults with an AUD who are receiving shelter-based treatment. Phase I will identify environmental (i.e., geolocation), cognitive, and behavioral antecedents of alcohol use over 4 weeks. Phase II will use this information to create a risk algorithm and tailored treatment messages that anticipate and intervene to prevent drinking. The resulting app will assess imminent risk of alcohol use after each EMA and will deliver relevant treatment messages that match a person's current risk factors. Phase III will test the feasibility, acceptability and preliminary efficacy of the app in a sample of 40 homeless adults with an AUD who receive the EMA plus treatment messages over 4 weeks. Drinking will be determined via self-report, supplemented by a transdermal alcohol sensor (i.e., SCRAM) worn by participants. This project will be the first to combine geolocation and psychosocial variables to identify real-time antecedents of drinking. If effective, this smartphone app could significantly improve treatment engagement, drinking outcomes, and quality of life among homeless adults with alcohol use disorders.

DETAILED DESCRIPTION:
An estimated 6.2% of US adults will be homeless at some point in their lifetime. Homeless adults have higher rates of disease, greater risk of interpersonal violence, shorter life expectancies, and disproportionately higher health care utilization and costs compared to housed individuals. A significant contributor to morbidity and mortality among homeless adults is the high prevalence of alcohol use. Approximately 33% of homeless adults have current alcohol dependence, a rate nearly 8 times that of the general population. Although shelter-based treatments are common, compliance is typically poor. Identifying factors that influence alcohol use would significantly improve the ability to develop effective interventions and engage homeless adults in treatment.

Relatively little is known about the environmental, cognitive, and behavioral antecedents of alcohol use in homeless adults. Like other subgroups, alcohol use has most often been examined using traditional lab/clinic based assessment methods that are not well suited to capturing the complicated street-level interactions experienced by most homeless adults. Traditional assessment methodologies may also provide biased and/or inaccurate estimates due to recall biases and errors in memory, particularly in this complicated population. Ecological momentary assessment (EMA), in which handheld devices (e.g., smartphones) are used to capture moment-to-moment experience, is currently the most accurate way to measure phenomena in natural settings. Additionally, recent technological advances have made it possible to collect continuous geolocation data alongside EMA. Researchers can now link environmental risks and protective factors to outcomes, without reliance on subjective reporting alone.

This pilot study will develop and test a "just-in-time" adaptive intervention to reduce alcohol use among homeless adults. Phase I will use smartphones and passive sensing to monitor geolocation, psychosocial variables (e.g., stress, urge to drink), and alcohol use in a group of 80 homeless adults enrolled in shelter-based treatment for an AUD. Phase II will use this information to create a risk algorithm and tailored treatment messages that anticipate and intervene to prevent alcohol use. Phase II will modify an existing app, previously validated for smoking cessation, to create the intervention. Phase III will pilot test the newly developed app for utility, satisfaction, and preliminary effectiveness in a group of 40 homeless adults with an AUD who are enrolled in shelter-based treatment. Alcohol consumption will be validated via a transdermal alcohol sensor (i.e., SCRAM) worn by participants in Phases I and III.

The central hypothesis is that alcohol use is strongly affected by moment-to-moment risk and protective factors. This study will be able to use EMAs to identify and automatically intervene during moments when people are at high risk for drinking. This hypothesis is based on preliminary findings among homeless, justice-involved, and socioeconomically disadvantaged safety-net hospital patients. If effective, this smartphone app could significantly improve treatment engagement, drinking outcomes, and quality of life among homeless adults with AUDs.

This project will:

1. Use EMA to identify environmental (i.e., geolocation), cognitive, and behavioral antecedents of alcohol use among 80 homeless adults with an AUD who are receiving shelter-based treatment.
2. Informed by Aim 1 findings, develop a "just-in-time" adaptive intervention to reduce alcohol use, including an alcohol use risk algorithm and corresponding theory-based treatment messages.
3. Examine feasibility, acceptability, and preliminary effectiveness of a just-in-time adaptive smartphone app among 40 homeless adults with an AUD who are receiving shelter-based treatment.

ELIGIBILITY:
Inclusion Criteria:

* Score ≥ 8 on the AUDIT
* Report consuming ≥ 1 drink of alcohol in the past week
* Receiving treatment at Metrocare;
* Willing and able to complete the baseline and follow-up visits;
* Score ≥ 4 on the REALM-SF, indicating > 6th grade English literacy level
* Score ≥ 24 on the Mini-Mental State Exam

Exclusion Criteria:

* Circulation problems, neuropathy, deep vein thrombosis, leg ulcers, tendonitis, diabetes, pregnancy, history of swelling or nickel or other metal allergies that would prohibit wearing the SCRAM ankle bracelet.
* Self-reported discomfort wearing an alcohol sensing bracelet for 4 weeks.
* Previously participated in Phase I (for Phase III recruitment).

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2019-02-14 (Actual); Primary Completion 2021-07-30 (Actual); Study Completion 2022-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott Walters, PhD, Principal Investigator — University of North Texas Health Science Center
Locations (1):
- Bridge Homeless Recovery Center, Dallas, Texas, United States

REFERENCES:
- [Result] Walters ST, Mun EY, Tan Z, Luningham JM, Hebert ET, Oliver JA, Businelle MS. Development and preliminary effectiveness of a smartphone-based, just-in-time adaptive intervention for adults with alcohol misuse who are experiencing homelessness. Alcohol Clin Exp Res. 2022 Sep;46(9):1732-1741. doi: 10.1111/acer.14908. Epub 2022 Aug 7. PMID 35869820
- [Result] Walters ST, Businelle MS, Suchting R, Li X, Hebert ET, Mun EY. Using machine learning to identify predictors of imminent drinking and create tailored messages for at-risk drinkers experiencing homelessness. J Subst Abuse Treat. 2021 Aug;127:108417. doi: 10.1016/j.jsat.2021.108417. Epub 2021 Apr 20. PMID 34134874
- [Result] Mun EY, Li X, Businelle MS, Hebert ET, Tan Z, Barnett NP, Walters ST. Ecological Momentary Assessment of Alcohol Consumption and Its Concordance with Transdermal Alcohol Detection and Timeline Follow-Back Self-report Among Adults Experiencing Homelessness. Alcohol Clin Exp Res. 2021 Apr;45(4):864-876. doi: 10.1111/acer.14571. Epub 2021 Mar 3. PMID 33583057
- [Result] Businelle MS, Walters ST, Mun EY, Kirchner TR, Hebert ET, Li X. Reducing Drinking Among People Experiencing Homelessness: Protocol for the Development and Testing of a Just-in-Time Adaptive Intervention. JMIR Res Protoc. 2020 Apr 16;9(4):e15610. doi: 10.2196/15610. PMID 32297874

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | EMA Only | EMA + App/Treatment Messages
Started | 78 | 41
Completed | 71 | 34
Not Completed | 7 | 7

BASELINE CHARACTERISTICS:
Population: Baseline reporting shows participants who completed the phone setup visit. For drinking outcomes, we limited the analysis to participants who had at least eight days of EMA reporting over the follow-up period. Because this pilot study aimed to examine the preliminary effectiveness of a new app, we deemed it necessary to have at least a seven-day exposure to the app (out of a maximum of 28 days) to reasonably test whether the app was efficacious.
Groups:
- Total: Total of all reporting groups
Arm/Group | EMA Only | EMA + App/Treatment Messages | Total
Number analyzed (Participants) | 78 | 41 | 119
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 78 | 41 | 119
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.6 (9.2) | 45.2 (11.5) | 46.1 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 8 | 20
  Male | 66 | 33 | 99
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 22 | 10 | 32
  White | 51 | 29 | 80
  More than one race | 2 | 2 | 4
  Unknown or Not Reported | 2 | 0 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 78 | 41 | 119

OUTCOME MEASURES:

1. Primary Outcome: Satisfaction With App Treatment Messages
Description: Satisfaction with app on self-reported questions at follow-up (1-5 scale where 1 = Not at all; and 5 = Extremely)
Time Frame: 4 weeks
Population: People who attended 4-week follow-up visit
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | EMA Only | EMA + App/Treatment Messages
Number analyzed (Participants) | 0 | 33
score on a scale
  How useful was the "Sober Tips" feature? |  | 3.9 (1.0)
  How helpful has the smart phone application been in helping you to reduce alcohol consumption? |  | 3.6 (1.1)
  Would you be interested in using this smart phone app in the future if needed? |  | 3.8 (1.5)
  How likely would you be to recommend this smart phone app to a friend? |  | 4.0 (1.4)

2. Secondary Outcome: Number of Drinking Days
Description: Number of drinking days (number of days with any self-reported drinking out of 28 days)
Time Frame: 4 weeks
Population: Participants available for analysis
Measure: Mean (Standard Deviation); unit: Number of drinking days
Arm/Group | EMA Only | EMA + App/Treatment Messages
Number analyzed (Participants) | 43 | 34
Number of drinking days | 13.9 (2.65) | 11.2 (2.60)

3. Secondary Outcome: Number of Heavy Drinking Days
Description: Number of drinking days (number of days with self-reported >4 drinks for men; >3 drinks for women out of 28 days)
Time Frame: 4 weeks
Population: Participants available for analysis
Measure: Mean (Standard Deviation); unit: Number of heavy drinking days
Arm/Group | EMA Only | EMA + App/Treatment Messages
Number analyzed (Participants) | 43 | 34
Number of heavy drinking days | 3.42 (1.78) | 3.64 (1.73)

ADVERSE EVENTS:
Time Frame: 4 weeks
Description: * Upon learning of an SAE or unanticipated AE, study staff will inform the local project manager as soon as possible (but within 48 hours of discovery).
  * The PIs review the Negative Event Incident Report and submit it to the IRBs and/or funder as required.
  * The PIs will ensure that SAEs and unanticipated AEs are followed until a final disposition of the adverse event is made.
  * The PIs will evaluate each SAE or unanticipated AE to determine whether it is related to the study.
Arm/Group | EMA Only | EMA + App/Treatment Messages
All-Cause Mortality (participants affected / at risk) | 0/78 | 0/41
Serious Adverse Events (participants affected / at risk) | 0/78 | 0/41
Other Adverse Events (participants affected / at risk) | 0/78 | 0/41

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-11-02): https://cdn.clinicaltrials.gov/large-docs/08/NCT03746808/Prot_SAP_000.pdf